CLINICAL TRIAL: NCT03953053
Title: Safety and Efficacy of FLACS With the FEMTO LDV Z8 Laser Compared to Conventional Cataract Surgery in Chinese Patients
Acronym: Z8CAT01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziemer Ophthalmic Systems AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FL5940-0001-CN
Record Dates: First submitted 2019-05-15; First posted 2019-05-16 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Cataract
Keywords: Femto Cataract Surgery
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FLACS Group (Experimental): Femto Laser treated (anterior Capsulotomy and Fragmentation of lens body before phaco emulification)
  Interventions: Device: Femtosecond Laser Assissted Cataract Surgery
- Manual Group (Active Comparator): Gold Standard Method with manual rhexis with pinzette and phaco emulsification
  Interventions: Device: Femtosecond Laser Assissted Cataract Surgery

INTERVENTIONS:
Device: Femtosecond Laser Assissted Cataract Surgery — During routine Catarct Surgery the Femtolaser cuts a ACCC (Anterior Continous Curvilinear Capsulotomy) into the lensbag and fragmentise the cataract affilited lens body

SUMMARY:
This trial will be designed as a multi-center randomized non-inferiority clinical trial to demonstrate safety and efficacy of the FEMTO LDV Z8 laser for cataract surgery in a Chinese population in China compared to the conventional technique.

DETAILED DESCRIPTION:
In this three center, prospective, interventional, randomized controlled study we aim to determine safety and efficacy of the FEMTO LDV Z8 laser as compared to conventional technique in Chinese patients diagnosed with cataract of any severity grade that are eligible to undergo cataract surgery with age 50 years and a maximum age of 80 years in China.

ELIGIBILITY:
Inclusion Criteria:

* Eligible to undergo cataract extraction by phacoemulsification with primary intraocular lens implantation
* Provision of signed and dated informed consent form
* Male or female, between 50 and 80 years of age (50 and 80 are included).
* IOL chosen for implantation a monofocal aspheric IOL of 6mm optic diameter
* Willing to comply with all study procedures and able to return for scheduled follow-up examinations
* Willing to adhere to the medication (to prevent inflammation and infection) regimen

Exclusion Criteria:

* Corneal disease or pathology, such as corneal scaring or opacity, that precludes transmission of laser wavelength or that distorts laser light
* Poorly dilating pupil or other defect of the pupil that prevents the iris from adequate retraction peripherally (e.g., intraoperative floppy iris syndrome)
* Glaucoma or ocular hypertension, pseudoexfoliation
* Corneal endothelial pathology where endothelial cell count is compromised (Fuchs endothelial dystrophy and others)
* Complicated cataract, such as traumatic, white, intumescent or posterior and anterior subcapsular cataracts
* Nystagmus or hemofacial spasm preventing placement of the patient interface
* Previous intraocular or corneal surgery of any kind, including any type of surgery for either refractive or therapeutic purposes in either eye
* Allergy to medications required in surgery, pre- and post-operative treatment
* History of lens or zonular instability
* Keratoconus or keratectasia
* Immune compromised or diagnosis of ophthalmic disease: ocular herpes zoster or simplex, lupus, collagenosis and other acute or chronic illnesses that increases the risk to the subject or confounds the outcomes of this study in the opinion of the study PI (Principal Investigator)
* Anterior chamber depth (ACD) < 1.5 mm or > 4.8 mm as measured from the corneal endothelium.
* Developmental disability or cognitive impairment that would make informed consent and the assessment of visual acuity impossible
* Concurrent participation in another ophthalmological clinical study

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-06-04 (Actual)

PRIMARY OUTCOMES:
Endothelial cell loss | 4 month
  To determine whether the FLACS with the FEMTO LDV Z8 laser is non-inferior to measured using the NSP 9900, KONAN MEDICAL, and calculated according to: postoperative endothelial cell loss = preoperative endothelial count - postoperative endothelial cell count

SECONDARY OUTCOMES:
Intra- and post- surgical complications | 4 month
  Diagnosis of Complications in combination with usual follow-up measures
Cumulative dissipated energy (CDE) | 4 month
  Recording of CDE on Phaco device
Ultrasound (US) total time | 4 month
  Record of US Energy applied
Estimated fluid usage (EFU) | 4 month
  Record of EFU
Corneal thickness (CCT) | 4 month
  Mesurement of the Central Corneal Thickness
Uncorrected distance visual acuity (UDVA) | 4 month
  Measurement of UDVA
Corrected distance visual acuity (CDVA) | 4 month
  Measurement of CDVA

CONTACTS AND LOCATIONS:
Overall Officials: A-Yong Yu, MD PHD Prof., Principal Investigator — The Eye Hospital of Wenzhou Medical University
Locations (1):
- Ziemer Ophthalmic Systems AG, Port, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou KJ, Huang Y, Wang Y, Pan AP, Shao X, Tu RX, Yu AY. Safety and efficacy of cataract surgery performed with a low-energy femtosecond laser compared with conventional phacoemulsification in Chinese patients: a randomized clinical trial. Eye Vis (Lond). 2023 Jul 2;10(1):31. doi: 10.1186/s40662-023-00347-0. PMID 37393278